CLINICAL TRIAL: NCT03759665
Title: Effects of N-Acetyl-L-Leucine on GM2 Gangliosidosis (Tay-Sachs and Sandhoff Disease): A Multinational, Multicenter, Open-label, Rater-blinded Phase II Study
Brief Title: N-Acetyl-L-Leucine for GM2 Gangliosidosis (Tay-Sachs and Sandhoff Disease)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IntraBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IB1001-202
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: GM2 Gangliosidosis; Tay-Sachs Disease; Sandhoff Disease
MeSH Terms: conditions — Gangliosidoses, GM2; Tay-Sachs Disease; Sandhoff Disease | interventions — IB1001; acetylleucine

STUDY DESIGN:
Intervention Model Description: In both the Parent Study and Extension Phase, patients will be assessed during three study phases: a baseline period (with or without a study run-in), a treatment period, and a washout period.
Who Masked: Outcomes Assessor
Masking Description: The primary evaluation of the Clinical Impression of Change in Severity (CI-CS; Primary Endpoint) will be performed by two independent neurologists whose assessments are based on videos of patient's performance on either the 9 Hole Peg Test of the Dominant Hand (9HPT-D) or the 8 Meter Walk Test (8MWT) taken at each visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with IB1001 (Experimental): Parent Study: 6-weeks treatment with IB1001 administered orally. Extension Phase: 1-year treatment with IB1001 administered orally.
  Patients ≥13 years old will receive a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old will receive weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg will take 2 g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg will take 3 g per day: 1 g in the morning, 1 g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg will take 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  Interventions: Drug: IB1001
- Post-Treatment Washout (No Intervention): After the Parent Study 6-week treatment period, and Extension Phase one-year treatment period, patients will enter a 6-week post-treatment washout period.

INTERVENTIONS:
Drug: IB1001 — IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  Other Names: N-Acetyl-L-Leucine
  Arms: Treatment with IB1001

SUMMARY:
This is a multinational, multicenter, open-label, rater-blinded prospective Phase II study which will assess the safety and efficacy of N-Acetyl-L-Leucine (IB1001) for the treatment of GM2 Gangliosidosis (Tay-Sachs and Sandhoff Disease).

There are two phases to this study: the Parent Study, and the Extension Phase.

The Parent Study evaluates the safety and efficacy of N-Acetyl-L-Leucine (IB1001) in the symptomatic treatment of GM2 Gangliosidosis (Tay-Sachs and Sandhoff Disease).

The Extension Phase evaluates the long-term safety and efficacy of IB1001 for the neuroprotective, disease-modifying treatment of GM2 Gangliosidosis. The Extension Phase was considered exploratory.

DETAILED DESCRIPTION:
In the Parent Study, Patients will be assessed during three study phases: a baseline period, a 6-week treatment period, and a 6-week post-treatment washout period. If within 6 weeks prior to the initial screening visit, a patient has received any of the prohibited medications defined in the eligibility criteria (irrespective of the preceding treatment duration) a wash-out study-run-in of 6 weeks is required prior to the first baseline assessment. All patients will receive the study drug during the treatment period. For each individual patient, the Parent Study lasts for approximately 3.5 - 4 months during which there are 6 visits to the study site.

This Extension Phase allows patients who have completed the Parent Study to, at the discretion of the Principal Investigator (PI), continue treatment with N-Acetyl-L-Leucine (IB1001). Patients will receive treatment with IB1001 for two one-year treatment periods, separated by a 6-week washout. All patients will receive the study drug during these two one-year treatment periods. For each individual patient, the Extension Phase lasts for approximately 25.5 months, during which there are 6 visits to the study site.

ELIGIBILITY:
Parent Study Inclusion Criteria

Individuals who meet all of the following criteria are eligible to participate in the study:

1. Written informed consent signed by the patient and/or their legal representative/ parent
2. Male or female aged ≥6 years in Europe OR ≥18 years in the United States with a confirmed diagnosis of GM2 Gangliosidosis ( i.e., clinical features and positive genetic test GM2-gangliosidosis caused by β-hexosaminidase deficiency resulting from mutations in the HEXA or HEXB genes) at the time of signing informed consent.
3. Females of childbearing potential, defined as a premenopausal female capable of becoming pregnant, will be included if they are either sexually inactive (sexually abstinent for 14 days prior to the first dose continuing through 28 days after the last dose) or using one of the following highly effective contraceptives (i.e. results in <1% failure rate when used consistently and correctly) 14 days prior to the first dose continuing through 28 days after the last dose:

   1. intrauterine device (IUD);
   2. surgical sterilization of the partner (vasectomy for 6 months minimum);
   3. combined (estrogen or progestogen containing) hormonal contraception associated with the inhibition of ovulation (either oral, intravaginal, or transdermal);
   4. progestogen-only hormonal contraception associated with the inhibition of ovulation (either oral, injectable, or implantable);
   5. intrauterine hormone-releasing system (IUS);
   6. bilateral tubal occlusion.
4. Females of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

   1. hysteroscopic sterilization;
   2. bilateral tubal ligation or bilateral salpingectomy;
   3. hysterectomy;
   4. bilateral oophorectomy;

   OR

   be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status. FSH analysis for postmenopausal women will be done at screening. FSH levels should be in the postmenopausal range as determined by the central laboratory.
5. Non-vasectomized male patient agrees to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study medication and the female partner agrees to comply with inclusion criteria 3 or 4. For a vasectomized male who has had his vasectomy 6 months or more prior to study start, it is required that they use a condom during sexual intercourse. A male who has been vasectomized less than 6 months prior to study start must follow the same restrictions as a non-vasectomized male.
6. If male, the patient agrees not to donate sperm from the first dose until 90 days after dosing.
7. Patients must fall within:

   a) A Scale for the Assessment and Rating of Ataxia (SARA) score of 5 ≤ X ≤ 33 points (out of 40) AND i. Within the 2-7 range (out of 0-8 range) of the Gait subtest of the SARA scale OR ii. Be able to perform the 9 Hole Peg Test with Dominant Hand (9HPT-D) (SCAFI subtest) in 20 ≤ X ≤150 seconds.
8. Weight ≥15 kg at screening.
9. Patients are willing to disclose their existing medications/therapies for (the symptoms) of GM2 Gangliosidosis, including those on the prohibited medication list. Non-prohibited medications/therapies (e.g. concomitant speech therapy, and physiotherapy) are permitted provided:

   1. The Investigator does not believe the medication/therapy will interfere with the study protocol/results
   2. Patients have been on a stable dose/duration and type of therapy for at least 6 weeks before Visit 1 (Baseline 1)
   3. Patients are willing to maintain a stable dose/do not change their therapy throughout the duration of the study.
10. An understanding of the implications of study participation, provided in the written patient information and informed consent by patients or their legal representative/parent, and demonstrates a willingness to comply with instructions and attend required study visits (for children this criterion will also be assessed in parents or appointed guardians).

Parent Study Exclusion Criteria

Individuals who meet any of the following criteria are not eligible to participate in the study:

1. Asymptomatic patients
2. Patient has clinical features of Tay-Sachs or Sandhoff disease, but a completely negative result on a previous genetic test for GM2 Gangliosidosis caused by β-hexosaminidase deficiency resulting from mutations in the HEXA or HEXB genes
3. Patients who have any of the following:

   1. Chronic diarrhea;
   2. Unexplained visual loss;
   3. Malignancies;
   4. Insulin-dependent diabetes mellitus.
   5. Known history of hypersensitivity to the N-Acetyl-Leucine (DL-, L-, D-) or derivatives.
   6. History of known hypersensitivity to excipients of Ora-Blend® (namely sucrose, sorbitol, cellulose, carboxymethylcellulose, xanthan gum, carrageenan, dimethicone, methylparaben, and potassium sorbate).
4. Simultaneous participation in another clinical study or participation in any clinical study involving administration of an investigational medicinal product (IMP; 'study drug') within 6 weeks prior to Visit 1.
5. Patients with a physical or psychiatric condition which, at the investigator's discretion, may put the patient at risk, may confound the study results, or may interfere with the patient's participation in the clinical study.
6. Known clinically-significant (at the discretion of the investigator) laboratories in hematology, coagulation, clinical chemistry, or urinalysis, including, but not limited to:

   1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5x upper limit of normal (ULN);
   2. Total bilirubin >1.5x ULN, unless Gilbert's syndrome is present in which case total bilirubin >2x ULN.
7. Known or persistent use, misuse, or dependency of medication, drugs, or alcohol.
8. Current or planned pregnancy or women who are breastfeeding.
9. Patients with severe vision or hearing impairment (that is not corrected by glasses or hearing aids) that, at the investigator's discretion, interferes with their ability to perform study assessments.
10. Patients who have been diagnosed with arthritis or other musculoskeletal disorders affecting joints, muscles, ligaments, and/or nerves that by themselves affects patient's mobility and, at the investigator's discretion, interferes with their ability to perform study assessments.
11. Patients unwilling and/or not able to undergo a 6-week washout period from any of the following prohibited medication prior to Visit 1 (Baseline 1) and remain without prohibited medication through Visit 6.

    1. Aminopyridines (including sustained-release form);
    2. N-Acetyl-DL-Leucine (e.g. Tanganil®);
    3. N-Acetyl-L-Leucine (prohibited if not provided as IMP);
    4. Riluzole;
    5. Gabapentin;
    6. Varenicline;
    7. Chlorzoxazone;
    8. Sulfasalazine;
    9. Rosuvastatin.

Extension Phase Inclusion Criteria

1. Completed Visit 6 of the IB1001-202 Parent Study
2. The Principal Investigator determines further treatment with IB1001 to be in the patient's best interest
3. Written informed consent signed by the patient and/or their legal representative/parent/ impartial witness for participation in the Extension Phase
4. Patients are willing to continue to remain without the following prohibited medication from Visit 6 throughout the duration of the Extension Phase:

Aminopyridines (including sustained-release form); b) N-Acetyl-DL-Leucine (e.g. Tanganil®); c) N-Acetyl-L-Leucine (prohibited if not provided as IMP); d) Riluzole; e) Gabapentin; f) Varenicline; g) Chlorzoxazone; h) Sulfasalazine; i) Rosuvastatin.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - University of California - Los Angeles, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone School of Medicine, New York, New York
- Germany (2):
  - University of Giessen, Giessen
  - Ludwig Maximilian University of Munich, München
- Bellvitge University Hospital, Barcelona, Spain
- United Kingdom (2):
  - Salford Trust, Salford, Greater Manchester
  - Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Derived] Martakis K, Claassen J, Gascon-Bayari J, Goldschagg N, Hahn A, Hassan A, Hennig A, Jones S, Kay R, Lau H, Perlman S, Sharma R, Schneider S, Bremova-Ertl T. Efficacy and Safety of N-Acetyl-l-Leucine in Children and Adults With GM2 Gangliosidoses. Neurology. 2023 Mar 7;100(10):e1072-e1083. doi: 10.1212/WNL.0000000000201660. Epub 2022 Dec 1. PMID 36456200
- [Derived] Churchill GC, Strupp M, Factor C, Bremova-Ertl T, Factor M, Patterson MC, Platt FM, Galione A. Acetylation turns leucine into a drug by membrane transporter switching. Sci Rep. 2021 Aug 4;11(1):15812. doi: 10.1038/s41598-021-95255-5. PMID 34349180
- [Derived] Fields T, Patterson M, Bremova-Ertl T, Belcher G, Billington I, Churchill GC, Davis W, Evans W, Flint S, Galione A, Granzer U, Greenfield J, Karl R, Kay R, Lewi D, Mathieson T, Meyer T, Pangonis D, Platt FM, Tsang L, Verburg C, Factor M, Strupp M. A master protocol to investigate a novel therapy acetyl-L-leucine for three ultra-rare neurodegenerative diseases: Niemann-Pick type C, the GM2 gangliosidoses, and ataxia telangiectasia. Trials. 2021 Jan 22;22(1):84. doi: 10.1186/s13063-020-05009-3. PMID 33482890

RESULTS

PARTICIPANT FLOW:
Groups:
- Parent Study: 6-weeks treatment with IB1001 administered orally. Patients ≥13 years old received a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took take 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults).
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period, patients entered a 6-week post-treatment washout period.
Period: Treatment With IB1001
Arm/Group | Parent Study
Started | 30
Completed | 27
Not Completed | 3
Period: Post-Treatment Washout
Arm/Group | Parent Study
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Parent Study: All patients were first dosed with IB1001.Therefore, the baseline characteristics of patients dosed in the first IB1001treatment period in the parent study constitute the baseline characteristics for the entire study.
Arm/Group | Parent Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 10
  United Kingdom | 1
  Germany | 18
  Spain | 1
Tay-Sachs vs. Sandhoff Patients [Number; unit: participants]
  Tay-Sachs | 27
  Sandhoff | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Impression of Change in Severity (CI-CS) [Fields et al 2021]
Description: The Clinical Impression of Change in Severity assessment will instruct the blinded rater to consider: compared to the first video, how has the severity of their performance on the 9 Hole Peg Test of the Dominant Hand (9HPT-D) or 8 Meter Walk Test (8MWT) changed (improved or worsened) in 6-weeks as observed in the second video? The Clinical Impression of Change in Severity is evaluated on a 7 point Likert scale (+3=significantly improved to -3= significantly worse).
  Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4)). Then, the mean change obtained in the post-treatment period was subtracted from the mean change obtained for the treatment with IB1001 period, with a positive value indicating an improvement in the treatment period compared to the post-treatment washout period.
Time Frame: (CI-CS comparing Baseline [Day 1] with IB1001 versus the end of 6-weeks treatment with IB1001 [approximately Day 42]) MINUS (CI-CS comparing the end of 6-weeks treatment with IB1001 [approximately Day 42] versus end of 6-weeks post-treatment washout);
Population: Modified Intention to Treat (mITT) Analysis Set is defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parent Study: 6-weeks treatment with IB1001administered orally. Patients ≥13 years old received a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period,patients entered a 6-week post-treatment washout period.
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale | 0.71 (2.09)
Statistical Analysis 1: Comparison: Parent Study; Test type: Superiority; p = 0.044, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = 0.75, 90% CI 2-sided [0.00 to 1.50]

2. Secondary Outcome: Key Secondary Endpoint: Individual Components of the CI-CS
Description: The Clinical Impression of Change in Severity assessment will instruct the blinded rater to consider: compared to the first video, how has the severity of their performance on the 9 Hole Peg Test of the Dominant Hand (9HPT-D) or 8 Meter Walk Test (8MWT) changed (improved or worsened) in 6-weeks as observed in the second video? The Clinical Impression of Change in Severity is evaluated on a 7 point Likert scale (+3=significantly improved to -3= significantly worse).
  Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4)).
Time Frame: Baseline to end of treatment with IB1001 (Parent Study 6-weeks treatment); End of treatment with IB1001 to the end of post 6-week treatment washout.
Population: Modified Intention to Treat (mITT) Analysis Set is defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 29 participants had values for the CI-CS analysis in the Treatment with IB1001 period and 27 participants in the Post-Treatment washout period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parent Study: 6-weeks treatment with IB1001 administered orally. Patients ≥13 years old received a total daily dose of 4 g/day (administered as 3 doses per day)
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period, patients entered a 6-week post-treatment washout period.
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment with IB1001 | 0.34 (1.59)
  Post-TreatmentWashout: number analyzed (Participants) | 27
  Post-TreatmentWashout | -0.36 (1.33)

3. Secondary Outcome: Key Secondary Endpoint: Change in Severity Based on Average CI-S
Description: The Change in Severity assessment will instruct the blinded rater to consider the severity of the patient at each visit.
  The Clinical Impression of Severity (CI-S)-assessment ranged from +3 ="normal not ill at all" to -3="among the most extremely ill patients ".
  Change values were calculated for each period, i.e. treatment with IB1001 (change between the baseline period (average for Visit 1 and Visit 2) and end of treatment period (average for Visit 3 and Visit 4)) and post-treatment washout (between end of treatment period (average for Visit 3 and Visit 4) and end of washout period (average for Visit 5 and Visit 6). Then, the mean change in the post-treatment period was subtracted from the mean change in the treatment with IB1001 period.
Time Frame: (CI-S comparing baseline period [average for Visit 1 and 2] and end of treatment period [average for Visit 3 and 4]) minus (change in CI-S between end of treatment period [average for Visit 3 and 4] and end of washout period [average for Visit 5 and 6]).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parent Study: 6-weeks treatment with IB1001 administered orally. Patients ≥13 years old received a total daily dose of 4 g/day (administered as 3 doses per day)
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine)is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period, patients entered a 6-week post-treatment washout period.
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale | 0.09 (0.71)
Statistical Analysis 1: Comparison: Parent Study; Test type: Superiority; p = 0.206, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = 0.13, 90% CI 2-sided [-0.13 to 0.25]

4. Secondary Outcome: Key Secondary Endpoint: CI-CS Score Reclassified on a 3-Point Scale
Description: The Clinical Impression of Change in Severity assessment will instruct the blinded rater to consider: compared to the first video, how has the severity of their performance on the 9 Hole Peg Test of the Dominant Hand (9HPT-D) or 8 Meter Walk Test (8MWT) changed (improved or worsened) in 6-weeks as observed in the second video? The Clinical Impression of Change in Severity is evaluated on a 7 point Likert scale (+3=significantly improved to -3= significantly worse).
  CI-CS scores <0 were reclassified as worsened (-1), CI-CS scores 0 remained classified as not changed (0), and CI-CS scores >0 were reclassified as improved (+1).
  When comparing Visit 4 versus Visit 2 and Visit 6 versus Visit 4, CI-CS scores <0 were reclassified as worsened (-1), CI-CS scores 0 remained classified as not changed (0), and CI-CS scores >0 were reclassified as improved (+1).
Time Frame: as for outcome 2
Population: The Modified Intention to Treat (mITT) analysis set was defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 29 participants had values for the CI-CS analysis in the Treatment with IB1001 period and 27 participants in the Post-Treatment washout period.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Study
Number analyzed (Participants) | 29
Participants
  Treatment with IB1001: -1 (Worsened) | 12
  Treatment with IB1001: 0 (No observable change) | 1
  Treatment with IB1001: +1 (Improved) | 16
  Post-treatment washout: number analyzed (Participants) | 27
  Post-treatment washout: -1 (Worsened) | 16
  Post-treatment washout: 0 (No observable change) | 3
  Post-treatment washout: +1 (Improved) | 8

5. Secondary Outcome: Key Secondary Endpoint: CI-CS Score for the Non-Primary Anchor Test
Description: as for outcome 2
Time Frame: CI-CS of the non-primary anchor test was evaluated, comparing the CI-CS of Visit 4 (end of treatment) versus Visit 2 (baseline) and of Visit 6 (end of washout) versus Visit 4 (end of treatment) as done for the primary anchor test.
Population: Modified Intention to Treat (mITT) Analysis Set is defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 22 participants had values for the CI-CS Score for the Non-Primary Anchor Test analysis in the Treatment with IB1001 period and 20 participants in the Post-Treatment washout period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment with IB1001: number analyzed (Participants) | 22
  Treatment with IB1001 | -0.30 (1.33)
  Post-treatment washout: number analyzed (Participants) | 20
  Post-treatment washout | 0.23 (1.43)

6. Secondary Outcome: Spinocerebellar Ataxia Functional Index (SCAFI) [Schmitz-Hübsch et al, 2008]
Description: Spinocerebellar Ataxia Functional Index (SCAFI) is composed of 8 Meter Walk Test, 9-Hole Peg Test of Dominant and Non-Dominant Hand (9HPT-D/9HPT-ND) (the 3 tests are timed assessments; each is done twice and values are averaged; the 8MWT and 9HPT-D and 9HPT-ND values are converted from times to rates, and the results expressed as a composite Z-score of each test relative to baseline) and the PATA rate (counted number how often a patient can repeat the syllables "PATA" within 10 seconds), a measure of speech performance. The scores of these 3 were transformed to Z-scores (=individual's average of both trials to perform the respective task -mean of study population at baseline) / SD of study population at baseline). A Z-score of 0 equates to the population mean at baseline. For all 3, higher Z-scores (above mean) mean better performance. The SCAFI total score was calculated as the arithmetic mean of the non-missing Z-scores for the 3. A higher total score means better performance.
Time Frame: Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4)).
Population: Modified Intention to Treat (mITT) Analysis Set is defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 26 participants had values for the SCAFI Total score analysis in the Treatment with IB1001 period and 25 participants in the Post-Treatment washout period
Measure: Mean (Standard Deviation); unit: Z-scores
Groups:
- Parent Study: 6-weeks treatment with IB1001 administered orally. Patients ≥13 years old in the United States received a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period, patients entered a 6-week post-treatment washout period.
Arm/Group | Parent Study
Number analyzed (Participants) | 29
Z-scores
  Treatment with IB1001: number analyzed (Participants) | 26
  Treatment with IB1001 | 0.0163 (0.2749)
  Post-treatment washout: number analyzed (Participants) | 25
  Post-treatment washout | -0.0080 (0.2420)
Statistical Analysis 1: Comparison: Parent Study; Treatment With IB1001; Test type: Superiority; p = 0.210, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = 0.0327, 90% CI 2-sided [-0.0327 to 0.1040]
Statistical Analysis 2: Comparison: Parent Study; Post-Treatment Washout; Test type: Superiority; p = 0.212, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = -0.0291, 90% CI 2-sided [-0.0863 to 0.0262]

7. Secondary Outcome: Scale for Assessment and Rating of Ataxia (SARA) Score [Schmitz-Hübsch Etal, 2006; Subramony, 2007]
Description: The Scale for Assessment and Rating of Ataxia has 8 items that are related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements, and heel-shin test. The range is 0-40 points, with a lower score representing neurological improvement and a higher score representing neurological worsening.
  Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4)).
Time Frame: Baseline to end of treatment with IB1001 (Parent Study Day 42); End of treatment with IB1001 to the end of post treatment washout
Population: The Modified Intention to Treat (mITT) analysis set was defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 28 participants had values for the SARA analysis in the Treatment with IB1001 period and 27 participants in the Post-Treatment washout period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parent Study: 6-weeks treatment with IB1001 administered orally. Patients ≥13 years old received a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period, patients entered a 6-week post-treatment washout period.
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment with IB1001: number analyzed (Participants) | 28
  Treatment with IB1001 | -1.41 (1.67)
  Post-treatment washout: number analyzed (Participants) | 27
  Post-treatment washout | 1.43 (2.08)
Statistical Analysis 1: Comparison: Parent Study; Treatment With IB1001; Test type: Superiority; p < 0.001, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = -1.25, 90% CI 2-sided [-1.75 to -0.75]
Statistical Analysis 2: Comparison: Parent Study; Post-Treatment Washout; Test type: Superiority; p = 0.001, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = 1.25, 90% CI 2-sided [0.50 to 2.00]

8. Secondary Outcome: EuroQuol- 5 Dimension (EQ-5D) Quality of Life Scale: Visual Analogue Scale (VAS)
Description: For posting, health-related quality of life based on the EQ-5D visual analogue scale (VAS) was presented as a secondary endpoint.
  EQ-5D VAS is a 0-100 scale where patients are asked to indicate their overall health, with a score of 0 indicating worst health and a score of 100indicating best health.
Time Frame: Baseline to end of treatment with IB1001 (Parent Study 6-week treatment): observed VAS values at visit 4; End of treatment with IB1001 to the end of post treatment washout: observed VAS values at visit 6.
Population: The Modified Intention to Treat (mITT) analysis set was defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 28 participants had values for the EQ-5D VAS analysis in the Treatment with IB1001 period and 27 participants in the Post-Treatment washout period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parent Study: 6-weeks treatment with IB1001 administered orally. Patients ≥13 years old received a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period ,patients entered a 6-week post-treatment washout period.
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment with IB1001: number analyzed (Participants) | 28
  Treatment with IB1001 | 71.3 (23.2)
  Post-Treatment Washout: number analyzed (Participants) | 27
  Post-Treatment Washout | 71.1 (21.2)

9. Secondary Outcome: Modified Disability Rating Scale (mDRS) [Iturriaga et al. 2006]
Description: Overall neurological status based on six domains (ambulation, manipulation,language, swallowing, seizures and ocular movements). The Modified Disability Rating Scale (mDRS) ranges from 0-24, where 0 is the best neurological status and 24 is the worst.
  Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4))
Time Frame: Baseline to end of treatment with IB1001 (Parent Study 6-weeks treatment); End of treatment with IB1001 to the end of post treatment washout.
Population: The Modified Intention to Treat (mITT) analysis set was defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 28 participants had values for the mDRS analysis in the Treatment with IB1001 period and 27 participants in the Post-Treatment washout period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment with IB1001: number analyzed (Participants) | 28
  Treatment with IB1001 | -0.030 (0.075)
  Post-Treatment Washout: number analyzed (Participants) | 27
  Post-Treatment Washout | 0.042 (0.058)
Statistical Analysis 1: Comparison: Parent Study; Treatment with IB1001; Test type: Superiority; p = 0.020, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = -0.031, 90% CI 2-sided [-0.063 to 0.000]
Statistical Analysis 2: Comparison: Parent Study; Post-Treatment Washout; Test type: Superiority; p < 0.001, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = 0.042, 90% CI 2-sided [0.021 to 0.063]

10. Secondary Outcome: Investigator's Clinical Global Impressions of Change (CGI-c)
Description: The Clinical Global Impression of Change assessed by the investigator is evaluated on a 7 point Likert scale ranging from 1='very much improved' to 7='very much worse'
  Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4)).
Time Frame: as for outcome 9
Population: The Modified Intention to Treat (mITT) analysis set was defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 28 participants had values for theInvestigator's CGI-C analysis in the Treatment with IB1001 period and 27 participants in the Post-Treatment washout period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parent Study: 6-weeks treatment with IB1001administered orally. Patients ≥13 years old received a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2g per day: 1 g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3g per day: 1 g in the morning, 1g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2 g in the morning, 1g in the afternoon and 1 g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
  After the 6-week treatment period, patients entered a 6-week post-treatment washout period.
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment with IB1001: number analyzed (Participants) | 28
  Treatment with IB1001 | 3.2 (1.0)
  Post-Treatment Washout: number analyzed (Participants) | 27
  Post-Treatment Washout | 4.9 (0.8)
Statistical Analysis 1: Comparison: Parent Study; Treatment With IB1001; Test type: Superiority; p < 0.001, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = 3.0, 90% CI 2-sided [3.0 to 3.5]
Statistical Analysis 2: Comparison: Parent Study; Post-Treatment Washout; Test type: Superiority; p < 0.001, 1-sided Wilcoxon signed-rank test; Hodges-Lehmann Estimator = 5.0, 90% CI 2-sided [4.5 to 5.0]

11. Secondary Outcome: Parent/Caregiver's Clinical Global Impression of Change (CGI-C)
Description: The Clinical Global Impression of Change assessed by the parent/caregiver is evaluated on a 7 point Likert scale ranging from 1='very much improved' to 7='very much worse'.
  Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4)).
Time Frame: Baseline to end of treatment with IB1001 (Parent Study 6-week treatment); End of treatment with IB1001 to the end of post treatment washout
Population: The Modified Intention to Treat (mITT) analysis set was defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 26 participants had values for the Parent/Caregiver's CGI-C analysis in the Treatment with IB1001 period and 25 participants in the Post-Treatment washout period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment With IB1001: number analyzed (Participants) | 26
  Treatment With IB1001 | 3.2 (1.2)
  Post-Treatment Washout: number analyzed (Participants) | 25
  Post-Treatment Washout | 4.8 (1.0)

12. Secondary Outcome: Patient's Clinical Global Impressions (CGI) if Able
Description: The Clinical Global Impression of Change assessed by the patient (if able) is evaluated on a 7 point Likert scale ranging from 1='very much improved' to 7='very much worse'.
  Change values were calculated for each period, i.e. treatment with IB1001 (comparing the end of treatment (Visit 4) with baseline (Visit 2)) and post-treatment washout (comparing the end of washout (Visit 6) with the end of treatment (Visit 4)).
Time Frame: as for outcome 9
Population: The Modified Intention to Treat (mITT) analysis set was defined as all patients who receive at least one dose of the study drug and with one video recording during the baseline period (Visit 1 or 2, or both) and treatment period (Visit 3 or Visit 4, or both). The overall mITT comprised 29 participants. Of these, 28 participants had values for the Patient's CGI if Able analysis in the Treatment with IB1001 period and 27 participants in the Post-Treatment washout period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Study
Number analyzed (Participants) | 29
score on a scale
  Treatment With IB1001: number analyzed (Participants) | 28
  Treatment With IB1001 | 3.0 (1.1)
  Post-Treatment Washout: number analyzed (Participants) | 27
  Post-Treatment Washout | 4.6 (1.2)

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form through to End of Study (Day 84, scheduled at 42 days post last IB1001dose).
Description: Adverse events (AEs) / serious adverse events (SAEs) consistent with the definition from ClinicalTrial.Gov. AEs/SAEs were collected in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-CGP).
Groups:
- Treatment With IB1001: Parent Study: 6-weeks treatment with IB1001 administered orally. Patients ≥13 years old in Europe and ≥18 years old in the United States received a total daily dose of 4 g/day (administered as 3 doses per day).
  Patients 6-12 years old received weight-tiered doses:
  * Patients aged 6-12 years weighing 15 to <25 kg took 2 g per day: 1g in the morning and 1 g in the evening.
  * Patients aged 6-12 years weighing 25 to <35 kg took 3 g per day: 1g in the morning, 1 g in the afternoon, and 1 g in the evening.
  * Patients aged 6-12 years weighing ≥35 kg took 4 g per day: 2g in the morning, 1 g in the afternoon and 1g in the evening (as per adults)
  IB1001: IB1001 (N-Acetyl-L-Leucine) is a modified amino-acid ester that is orally administered.
- Post-Treatment Washout: After the Parent Study 6-week treatment period, patients entered a 6-week post-treatment washout period.
Arm/Group | Treatment With IB1001 | Post-Treatment Washout
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/30
Other Adverse Events (participants affected / at risk) | 17/30 | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With IB1001 (N=30) | Post-Treatment Washout (N=30)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — The patient experienced a fracture of lumbar vertebrae due to a fall. The patient had recurrent falls in the medical history, as a symptom of Tay-Sachs disease and the investigator considered the event not related to study medication.
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — The patient experienced a fracture of lumbar vertebrae due to a fall. The patient had recurrent falls in the medical history, as a symptom of Tay-Sachs disease and the investigator considered the event not related to study medication.
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) — The patient suffered from concomitant bipolar disorder which deteriorated. The investigator judged the event not related to study medication.
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) — The patient suffered from concomitant bipolar disorder which deteriorated. The investigator judged the event not related to study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With IB1001 (N=30) | Post-Treatment Washout (N=30)
Fall (Injury, poisoning and procedural complications) | 7 (10) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Tremor (Nervous system disorders) | 4 (4) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was ongoing during the COVID-19 pandemic, and the conduct of this study was impacted by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03759665/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03759665/SAP_002.pdf